CLINICAL TRIAL: NCT05004558
Title: Effects of a 24-week Remote-based Resistance Training Program on Parameters of the Metabolic Syndrome, Cognitive Function, and Quality of Life in Older Adults Living With Mild Cognitive Impairment and Alzheimer's Disease and/or a Related Dementia
Brief Title: Effects of Remote-based Resistance Training on Cardiometabolic Risk Factors, Cognitive Function, and Quality of Life in Adults Living With Alzheimer's Disease and/or Related Dementias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Drexel University (Other)
Collaborators: Mercy Health (Other)
Responsible Party: Principal Investigator, Michael Bruneau, Assistant Professor, Drexel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THMA 2021-21
Record Dates: First submitted 2021-05-21; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Dementia; Alzheimer Disease; Dementia, Vascular; Lewy Body Disease; Frontotemporal Dementia; Mild Cognitive Impairment; Aging; Hypertension; Obesity, Abdominal; Obesity; Body Weight; Blood Pressure; Blood Glucose, High; Blood Glucose, Low; Dyslipidemias; Quality of Life; Cognitive Impairment
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Lewy Body Disease; Frontotemporal Dementia; Cognitive Dysfunction; Hypertension; Obesity, Abdominal; Obesity; Body Weight; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote-based Resistance Exercise Training (Experimental): All participants enrolled in the trial will receive supervised remote-based resistance exercise training. The exercises will be performed with the use of Therabands and will include 8-10 exercises performed for 1 set of 15 repetitions, performed 3 days per week for 24 weeks.
  Interventions: Other: Remote-based Resistance Exercise Training

INTERVENTIONS:
Other: Remote-based Resistance Exercise Training — All participants enrolled in the trial will receive supervised remote-based resistance exercise training. The exercises will be performed with the use of Therabands and will include 8-10 exercises performed for 1 set of 15 repetitions, performed 3 days per week for 24 weeks.

SUMMARY:
The investigators aim to study the effects of a 24-week remote-based resistance exercise training program on cardiovascular disease risk factors, cognitive function, and quality of life in older adults living with mild cognitive impairment or Alzheimer's Disease and/or a related dementia. Data for this study will be collected at the beginning, middle, and end of the resistance training program. Participants of this study will receive a baseline health-fitness assessment at the beginning of the study. Measurements of resting blood pressure, fasting blood glucose and lipids, waist and hip circumferences, height and weight, cognitive function and quality of life will be collected at the health-fitness assessment. Participants will then receive supervised remote-based resistance exercise training with Therabands, 3 days per week for 12 weeks before receiving a second 12-week health-fitness assessment in the middle of the intervention. Participants will then receive 12 additional weeks of supervised remote-based resistance exercise training with Therabands, 3 days per week for 12 weeks before receiving a third 24-week health fitness assessment at the end of the study.

DETAILED DESCRIPTION:
The investigators aim to study the effects of a 24-week remote-based resistance exercise training program on cardiovascular disease risk factors, cognitive function, and quality of life in older adults living with mild cognitive impairment or Alzheimer's Disease and/or a related dementia. Data for this study will be collected at the beginning, middle, and end of the resistance training program. Measurements of resting blood pressure will be collected with an automated blood pressure monitor. Fasting blood glucose and lipids will be retrieved from the electronic medical record or from a finger stick. Waist and hip circumferences will be collected with a tape measure. Height and weight will be collected with a physician scale. Cognitive function and quality of life will be collected from interviews using the Montreal Cognitive Assessment and Short-Form (36) Health Survey. All data collected from this study will be de-identified using the "Safe-Harbor" method, which minimizes exposure of personal health information by providing each participant with a unique participant-ID and only providing access to those who are listed and approved for access privileges. Data collected for this study will also be stored on an encrypted and password- protected hard drive, and data analyzed will be performed with the Statistical Package for the Social Sciences using analyses of covariance.

When participants are enrolled in the study, he/she will be grouped on the basis of their cognitive function status from the Montreal Cognitive Assessment. All participants will then receive supervised remote-based resistance exercise training with Therabands, 3 days per week for 24 weeks. The risks of participating in exercise programs are minimal. Some of the possible risks of participating in resistance exercise include becoming tired and/or experiencing delayed onset muscle soreness, leg cramping, or muscle strain from performing resistance exercise. There are several benefits from engaging in resistance exercise programs. Participants of this study will receive health-fitness assessment at the beginning, middle, and end of the study, and as such, will benefit from being made aware of their cardiovascular disease risk factors, cognitive function, and quality of life. Other possible benefits from participation in the resistance exercise program may include improvements in muscular size and strength and/or activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* Sedentary or not meeting the current physical activity guidelines of at least 150 minutes of moderate-to-vigorous physical activity per week
* Live with or have a primary in-home caregiver or legal representative who can be physically present during the remote-based exercise sessions
* Have access to a computer, tablet, or smartphone with internet and webcam access for the HIPAA compliant virtual Zoom meetings.

Exclusion Criteria:

* Younger than 55 years of age
* Accustomed to resistance exercise training during the previous year
* Live with known or suggestive uncontrolled cardiovascular, metabolic, and/or renal disease
* Live with musculoskeletal injury that precludes their ability to perform remote-based, resistance exercise training

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Resting systolic blood pressure, measured in mmHg from 0 and above with higher numbers indicating higher blood pressure | Baseline
  Resting systolic blood pressure will be measured with an automated blood pressure device, measured in mmHg from 0 and above with higher numbers indicating higher blood pressure
Resting systolic blood pressure, measured in mmHg from 0 and above with higher numbers indicating higher blood pressure | 12 weeks
  Resting systolic blood pressure will be measured with an automated blood pressure device, measured in mmHg from 0 and above with higher numbers indicating higher blood pressure
Resting systolic blood pressure, measured in mmHg from 0 and above with higher numbers indicating higher blood pressure | 24 weeks
  Resting systolic blood pressure will be measured with an automated blood pressure device, measured in mmHg from 0 and above with higher numbers indicating higher blood pressure
Resting diastolic blood pressure, measured in mmHg from 0 and above with higher numbers indicating higher blood pressure | Baseline
  Resting diastolic blood pressure will be measured with an automated blood pressure device, measured in mmHg from 0 and above with higher numbers indicating higher blood pressure
Resting diastolic blood pressure, measured in mmHg from 0 and above with higher numbers indicating higher blood pressure | 12 weeks
  Resting diastolic blood pressure will be measured with an automated blood pressure device, measured in mmHg from 0 and above with higher numbers indicating higher blood pressure
Resting diastolic blood pressure, measured in mmHg from 0 and above with higher numbers indicating higher blood pressure | 24 weeks
  Resting diastolic blood pressure will be measured with an automated blood pressure device, measured in mmHg from 0 and above with higher numbers indicating higher blood pressure
Height, red with a stadiometer in inches from 0 and above with higher numbers indicating taller height | Baseline
  Height will be measured with a stadiometer in inches from 0 and above with higher numbers indicating taller height
Height, red with a stadiometer in inches from 0 and above with higher numbers indicating taller height | 12 weeks
  Height will be measured with a stadiometer in inches from 0 and above with higher numbers indicating taller height
Height, red with a stadiometer in inches from 0 and above with higher numbers indicating taller height | 24 weeks
  Height will be measured with a stadiometer in inches from 0 and above with higher numbers indicating taller height
Weight, ured with a physican scale in pounds from 0 and above with higher numbers indicating heavier weight | Baseline
  Weight will be measured with a physican scale in pounds from 0 and above with higher numbers indicating heavier weight
Weight, ured with a physican scale in pounds from 0 and above with higher numbers indicating heavier weight | 12 weeks
  Weight will be measured with a physican scale in pounds from 0 and above with higher numbers indicating heavier weight
Weight, ured with a physican scale in pounds from 0 and above with higher numbers indicating heavier weight | 24 weeks
  Weight will be measured with a physican scale in pounds from 0 and above with higher numbers indicating heavier weight
Body mass index, measured in meters squared, from 0 and above wiith larger values indicating a higher body mass index | Baseline
  Body mass index will be measured as the weight measured in kilograms divided by the height measured in meters squared, from 0 and above wiith larger values indicating a higher body mass index
Body mass index, measured in meters squared, from 0 and above wiith larger values indicating a higher body mass index | 12 weeks
  Body mass index will be measured as the weight measured in kilograms divided by the height measured in meters squared, from 0 and above wiith larger values indicating a higher body mass index
Body mass index, measured in meters squared, from 0 and above wiith larger values indicating a higher body mass index | 24 weeks
  Body mass index will be measured as the weight measured in kilograms divided by the height measured in meters squared, from 0 and above wiith larger values indicating a higher body mass index
Waist circumference, red in inches with a Gulick tape measure from 0 and above with higher numbers indicating a larger waist circumference | Baseline
  Waist circumference will be measured in inches with a Gulick tape measure from 0 and above with higher numbers indicating a larger waist circumference
Waist circumference, red in inches with a Gulick tape measure from 0 and above with higher numbers indicating a larger waist circumference | 12 weeks
  Waist circumference will be measured in inches with a Gulick tape measure from 0 and above with higher numbers indicating a larger waist circumference
Waist circumference, red in inches with a Gulick tape measure from 0 and above with higher numbers indicating a larger waist circumference | 24 weeks
  Waist circumference will be measured in inches with a Gulick tape measure from 0 and above with higher numbers indicating a larger waist circumference
Hip circumference, sured in inches with a Gulick tape measure from 0 and above with higher numbers indicating a larger waist circumference | Baseline
  Hip circumference will be measured in inches with a Gulick tape measure from 0 and above with higher numbers indicating a larger waist circumference
Hip circumference, sured in inches with a Gulick tape measure from 0 and above with higher numbers indicating a larger waist circumference | 12 weeks
  Hip circumference will be measured in inches with a Gulick tape measure from 0 and above with higher numbers indicating a larger waist circumference
Hip circumference, sured in inches with a Gulick tape measure from 0 and above with higher numbers indicating a larger waist circumference | 24 weeks
  Hip circumference will be measured in inches with a Gulick tape measure from 0 and above with higher numbers indicating a larger waist circumference
Blood glucose, measured in mg/dL from 0 and above with larger values indicating a higher blood glucose concentration | Baseline
  Blood glucose will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher blood glucose concentration
Blood glucose, measured in mg/dL from 0 and above with larger values indicating a higher blood glucose concentration | 12 weeks
  Blood glucose will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher blood glucose concentration
Blood glucose, measured in mg/dL from 0 and above with larger values indicating a higher blood glucose concentration | 24 weeks
  Blood glucose will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher blood glucose concentration
High density lipoprotein cholesterol, ed in mg/dL from 0 and above with larger values indicating a higher high density lipoprotein concentrations, a desirable finding | Baseline
  High density lipoprotein cholesterol will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher high density lipoprotein concentrations, a desirable finding
High density lipoprotein cholesterol, ed in mg/dL from 0 and above with larger values indicating a higher high density lipoprotein concentrations, a desirable finding | 12 weeks
  High density lipoprotein cholesterol will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher high density lipoprotein concentrations, a desirable finding
High density lipoprotein cholesterol, ed in mg/dL from 0 and above with larger values indicating a higher high density lipoprotein concentrations, a desirable finding | 24 weeks
  High density lipoprotein cholesterol will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher high density lipoprotein concentrations, a desirable finding
Low density lipoprotein cholesterol, measured in mg/dL from 0 and above with larger values indicating a higher low density lipoprotein concentrations, an undesirable finding | Baseline
  Low density lipoprotein cholesterol will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher low density lipoprotein concentrations, an undesirable finding
Low density lipoprotein cholesterol, measured in mg/dL from 0 and above with larger values indicating a higher low density lipoprotein concentrations, an undesirable finding | 12 weeks
  Low density lipoprotein cholesterol will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher low density lipoprotein concentrations, an undesirable finding
Low density lipoprotein cholesterol, measured in mg/dL from 0 and above with larger values indicating a higher low density lipoprotein concentrations, an undesirable finding | 24 weeks
  Low density lipoprotein cholesterol will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher low density lipoprotein concentrations, an undesirable finding
Triglycerides, measured in mg/dL from 0 and above with larger values indicating a higher triglyceride concentrations, an undesirable finding | Baseline
  Triglycerides will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher triglyceride concentrations, an undesirable finding
Triglycerides, measured in mg/dL from 0 and above with larger values indicating a higher triglyceride concentrations, an undesirable finding | 12 weeks
  Triglycerides will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher triglyceride concentrations, an undesirable finding
Triglycerides, measured in mg/dL from 0 and above with larger values indicating a higher triglyceride concentrations, an undesirable finding | 24 weeks
  Triglycerides will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher triglyceride concentrations, an undesirable finding
Total cholesterol, measured in mg/dL from 0 and above with larger values indicating a higher total cholesterol concentrations, an undesirable finding | Baseline
  Total cholesterol will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher total cholesterol concentrations, an undesirable finding
Total cholesterol, measured in mg/dL from 0 and above with larger values indicating a higher total cholesterol concentrations, an undesirable finding | 12 weeks
  Total cholesterol will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher total cholesterol concentrations, an undesirable finding
Total cholesterol, measured in mg/dL from 0 and above with larger values indicating a higher total cholesterol concentrations, an undesirable finding | 24 weeks
  Total cholesterol will be measured with a Cholestech LDX analyzer via finger sticking, measured in mg/dL from 0 and above with larger values indicating a higher total cholesterol concentrations, an undesirable finding

SECONDARY OUTCOMES:
Cognitive Function as Measured by the Montreal Cognitive Assessment | Baseline
  Cognitive function will be assessed with the Montreal Cognitive Assessment Screen, measured from 0 to 30 with higher scores indicating better cognitive function
Cognitive Function as Measured by the Montreal Cognitive Assessment | 12 weeks
  Cognitive function will be assessed with the Montreal Cognitive Assessment Screen, measured from 0 to 30 with higher scores indicating better cognitive function
Cognitive Function as Measured by the Montreal Cognitive Assessment | 24 weeks
  Cognitive function will be assessed with the Montreal Cognitive Assessment Screen, measured from 0 to 30 with higher scores indicating better cognitive function
Quality of Life as measured by the Short-Form (36) Health Survey | Baseline
  Quality of life will be assessed with the Short-Form (36) Health Survey, measured from 0 to 100 with higher scores indicating better quality of life
Quality of Life as measured by the Short-Form (36) Health Survey | 12 weeks
  Quality of life will be assessed with the Short-Form (36) Health Survey, measured from 0 to 100 with higher scores indicating better quality of life
Quality of Life as measured by the Short-Form (36) Health Survey | 24 weeks
  Quality of life will be assessed with the Short-Form (36) Health Survey, measured from 0 to 100 with higher scores indicating better quality of life

IPD SHARING:
Plan to Share IPD: No